CLINICAL TRIAL: NCT05754593
Title: Study of Ovarian Reserve Concerning Patients With Multiple Sclerosis, Compared to a Control Group
Brief Title: Study of Ovarian Reserve Concerning Patients With Multiple Sclerosis (MS), Compared to a Control Group
Acronym: FEMINISEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/27
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; ovarian reserve; fertility; auto-immunity
MeSH Terms: conditions — Multiple Sclerosis | interventions — Anti-Mullerian Hormone; Floors and Floorcoverings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS patients (Experimental): Diagnosis of multiple sclerosis based on McDonald Criteria 2017
  Interventions: Biological: Anti-Mullerian hormone (AMH) level; Other: Antral follicle count (AFC); Other: Clinical assessment
- Controls (Active Comparator): Healthy controls
  Interventions: Biological: Anti-Mullerian hormone (AMH) level; Other: Antral follicle count (AFC)

INTERVENTIONS:
Biological: Anti-Mullerian hormone (AMH) level — Measure of Anti-Mullerian hormone (AMH) level by blood sample
Other: Antral follicle count (AFC) — Measure of Antral follicle count (AFC) by ultrasound imaging
Other: Clinical assessment — MS history and MS treatments and Expanded Disability Status Scale (EDSS) score will be recorded
  Arms: MS patients

SUMMARY:
The investigators want to evaluate ovarian reserve concerning patients with multiple sclerosis, compared to a control group of healthy women. This study will include women from 25 to 35 years old.

DETAILED DESCRIPTION:
Multiple sclerosis is an inflammatory disease of central nervous system, with a prevalence rate in France of 1 case/1000 subjects. The average age at diagnosis is 30 years old and it affects especially women, with a sex ratio of 3 women for 1 men. Multiples sclerosis concerns women at a moment when fertility is a main issue.

Few studies suggest that there is an negative impact of multiple sclerosis on ovarian reserve, with a combined mechanism ( inflammatory and autoimmune mechanism). The investigators can hypothesize that patients with multiple sclerosis are more predisposed to have primary ovarian insufficiency.

Ovarian reserve is evaluated by Anti-Mullerian Hormone (AMH) dosage and antral follicle count (AFC) by ultrasound imaging.AMH levels can be measured at every moment of the menstrual cycle whereas AFC is preferentially performed between the second and the eighth day of the menstrual cycle. The combined use of this two markers is well known to be correlated with ovarian reserve. Only a few studies have evaluated ovarian reserve in patients with multiple sclerosis. Besides, there is only a few number of participants and results are contradictory. A decrease of ovarian reserve identified among patients with multiple sclerosis could lead to an orientation in a fertility preservation center.

This project is a monocentric study realized at Pellegrin Hospital - Bordeaux. Patients with multiple sclerosis belong to a cohort of the neurology center. Healthy women come from a volunteer base contacted by email.The two groups are matched thanks to answers of a short questionnaire.Measure of AMH level is performed at pellegrin Hospital at the medical laboratory. Ultrasound imaging is performed by the center of women imagery at Pellegrin Hospital. Results are communicated by teleconsultation two months later. If there is an anormal result, a specific appointment will be organized with a gynecologist.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive women between 25 and 35 years old ;
* MS Patient : Diagnosis of multiple sclerosis based on McDonald Criteria 2017;
* French-speaking, without comprehension disorders ;
* being affiliated to health insurance ;
* Willing to participate and to sign informed consent.

Exclusion Criteria:

* History of ovarian surgery (cystectomy, annexectomy) ;
* Turner Syndrome ;
* fragile X messenger ribonucleoprotein 1 (FMR1) premutation ;
* Endometriosis with a risk of ovarian reserve alteration ;
* History of chemotherapy or pelvic radiotherapy ;
* Pregnant or breastfeeding women ;
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measure of Anti-Mullerian hormone (AMH) level by blood sample to compare ovarian reserve between patients with multiple sclerosis versus healthy controls from 25 to 35 years old. | At baseline (day 0)

SECONDARY OUTCOMES:
Measure of Antral follicle count (AFC) by ultrasound imaging to compare ovarian reserve between patients with multiple sclerosis versus healthy controls from 25 to 35 years old. | At baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BERNARD, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BERNARD, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de neurologie, Bordeaux, France